CLINICAL TRIAL: NCT07299682
Title: Facilitating Effective Eating With DoddleBags: A Single-Arm Acceptability Study Of DoddleBags to Assess Impact on Self Feeding Behaviours in a Huntington's Disease Population
Acronym: FEEDhd
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: FHS 23-24.95; 342883 (Other: HRA)
Record Dates: First submitted 2025-01-14; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Huntington's Disease (HD)

STUDY DESIGN:
Intervention Model Description: participants will provide baseline measurements for a defined period before all moving onto the intervention and providing further measurements after a second defined period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will undergo a pre-intervention semi-structured interview with the research after completing their ICF, they will also be asked to complete the questionnaire battery. Participants, with the aid of carers if appropriate, will then be asked to complete a food diary for one week to provide a baseline of their daily experiences. After this baseline week, participants will be asked to use the DoddleBags products in the preparation and execution of as many mealtimes as they reasonably can, while completing the food diaries for a further 11 weeks.
  Interventions: Device: DoddleBags

INTERVENTIONS:
Device: DoddleBags — DoddleBags are reusable flexible pouches that can be used as a feeding aid when filled with pureed textured food. They can be used with the included anti-choking cap or a spoon attachment as pictured. They are bisphenol A (BPA) free, leak proof and microwave and dishwasher safe.

SUMMARY:
Primary Objectives

* To assess the acceptability of using the DoddleBags feeding aid in people with HD, by using a food diary to track food intake and using semi-structured interviews to ask questions about how easy or difficult it was to use a DoddleBag for each meal compared to not using one, and learn more about the impact of using DoddleBags on self-feeding behaviours.
* To review the impact of using DoddleBags during mealtimes on the weight and BMI of each participant.
* To review the impact of using DoddleBags during mealtimes on episodes of choking of each participant.

Secondary Objectives

* To evaluate the impact of using DoddleBags on participants' attitudes towards mealtimes and eating, using a short battery of mood and eating questionnaires.
* To measure how incorporating DoddleBags into mealtimes affects participants' perceived quality of life, using a short battery of mood and eating questionnaires.
* To assess the acceptability of the short battery of mood and eating questionnaires within a population of people with HD.

DETAILED DESCRIPTION:
Study Procedure

* Design: Participants will be interviewed, complete questionnaires and use a food diary for a week to establish a baseline. Participants will then complete a food diary while using the DoddleBags for 11 weeks before completing the questionnaires and being interviewed again.
* Methods of data collection: The study makes use of a small battery of mood and eating questionnaires, as well as two semi-structured interviews and a food diary. The following questionnaires are proposed to form the battery:

  * Adult Eating Behaviours Questionnaire (AEB-Q)
  * Eating Attitude Test (EAT-26)
  * HD Quality of Life Scale (HDQoL)
  * HD-specific Eating Questionnaire (HD-EAT)
* Procedure: Participants will undergo a pre-intervention semi-structured interview with the research after completing the participants' ICF, participants will also be asked to complete the questionnaire battery. Participants, with the aid of carers if appropriate, will then be asked to complete a food diary for one week to provide a baseline of the participants' daily experiences. After this baseline week, participants will be asked to use the DoddleBags products in the preparation and execution of as many mealtimes as the participant reasonably can, while completing the food diaries for a further 11 weeks.

After both 1 and 4 weeks of using the DoddleBags the study team will contact the participants to check in with how the participants are finding incorporating the DoddleBags into mealtimes. As with every contact, it should be established that the participant is still happy to participate in the study and as part of the researchers' duty of care, researchers should explore if participants would like to withdraw from the study if the participant strongly believes the participant is receiving no significant benefits from the DoddleBags.

The post-intervention semi-structured interview and questionnaire battery will be completed in a study visit arranged as soon as reasonably possible, and ideally within the following week after the 11 week intervention period, to ensure the participants experiences are still fresh. After this the participants will be debriefed and participation will be considered complete.

• Analysis: The semi-structured interviews will be transcribed and fed into NVivo, software designed to facilitate thematic analysis. the researchers will conduct a reflexive thematic analysis on the transcripts to identify commonalities between the responses of participants both before and after the intervention. The AEBQ, HD-EAT, and HDQoL are quantitative measures, so the researchers will use a variety of explorative quantitative analyses to analysis the pre/post-intervention differences.

End of Study The study will be closed to recruitment after completion of informed consent for the final participant. The study team anticipates that participant involvement in the study will last around 12-13 weeks depending on how quickly the post-intervention semi-structured interview can be arranged at a convenient time for the participant. The study will be considered complete as a concept upon publication and submission of study results.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 or over at the time of recruitment.

Genetic confirmation of the HD gene expansion, defined as a CAG repeat length of ≥40 CAG repeats on the long allele.

Chorea, uncontrollable bodily movements, to the extent that it, in the opinion of the participant, inhibits normal or typical use of an eating utensil such as a fork or spoon.

AND/OR Cognitive issues that make it impractical for the participant to engage in self-feeding behaviours in a safe and effective manner, perhaps but not necessarily requiring the input of a carer or companion to feed the participant.

Exclusion Criteria:

Failing to meet the inclusion criteria.

The presence of a pre-existing neurological or movement disorder that could mimic, mask, or otherwise occlude the symptoms of Huntington's Disease.

Current use of DoddleBags as a feeding aid outside of this research.

Ability to regularly self-feed in a safe and effective manner rendering the integration of DoddleBags into one's lifestyle moot.

Use of a mandated/recommended diet that would be incompatible with DoddleBags, such as mandated use of non-pureed or non-soft foods.

Inability or unwillingness to engage with any specific aspects of the research, including completion of the food diaries, interviews or questionnaires, as well as being unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability | From enrollment to the end of treatment at 12 weeks.
  To assess the feasibility of using the DoddleBags feeding aid in people with HD, by using semi-structured interviews to ask questions about how easy or difficult it was to use a DoddleBag for each meal compared to not using one, and learn more about the impact of using DoddleBags on self-feeding behaviours.

SECONDARY OUTCOMES:
Attitudes Towards Mealtimes | From enrollment to the end of treatment at 12 weeks.
  To evaluate the impact of using DoddleBags on participants' attitudes towards mealtimes and eating, using the Eating Attitudes Test questionnaire.
Perceived Quality of Life | From enrollment to the end of treatment at 12 weeks.
  To measure how incorporating DoddleBags into mealtimes affects participants' perceived quality of life, using the Huntington's Disease Quality of Life questionnaire (HDQoL).

CONTACTS AND LOCATIONS:
Locations (7):
- United Kingdom (7):
  - Cambridge University Hospitals, Cambridge
  - Cardiff University, Cardiff
  - NHS Greater Glasgow & Clyde, Glasgow
  - Leeds Teaching Hospitals, Leeds
  - Leicestershire Partnership NHS Trust, Leicester
  - Walton Centre NHST, Liverpool
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No